CLINICAL TRIAL: NCT05489484
Title: Performance and Safety Evaluation of Type I Collagen (MD-Shoulder Collagen Medical Device) in the Treatment of Rotator Cuff Syndrome ''ROPIRAMED PILOT STUDY''
Brief Title: Performance and Safety Evaluation of MD-Shoulder Collagen Medical Device in the Treatment of Rotator Cuff Syndrome
Acronym: ROPIRAMED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guna S.p.a (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDG2021184
Record Dates: First submitted 2022-07-05; First posted 2022-08-05 (Actual); Results first posted 2025-07-08 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Rotator Cuff Tendinitis; Syndrome Rotator Cuff; Tendinopathy; Tendinoses, Rotator Cuff; Rotator Cuff Injuries
Keywords: Collagen Type I; MD-Shoulder Collagen Medical Device; Shoulder; Constant Murley Score; American Shoulder and Elbow Surgeons; Numeric Rating Scale; Simply Shoulder Test; Range of Motion
MeSH Terms: conditions — Rotator Cuff Injuries; Tendinopathy; Osteogenesis Imperfecta, Type IV

STUDY DESIGN:
Intervention Model Description: one sample study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MD-Shoulder Medical Device (Experimental): MD-Shoulder Medical Device type I collagen based
  Interventions: Device: MD-Shoulder Collagen Medical Device

INTERVENTIONS:
Device: MD-Shoulder Collagen Medical Device — Only one experimental group is scheduled by the Investigation Plan to be treated with 2-mL volume ultrasound-guided infiltrations of MD-Shoulder Collagen Medical Device (GUNA, Milan-Italy).
  Subjects will be treated with number one ultrasound-guided infiltration at the time of enrollment, 2 weeks after enrollment, and 4 weeks after enrollment.
  Intra-articular infiltrations will be performed with 5cc syringes and 22-gauge needles.
  MD-Shoulder Collagen Medical Device will be infiltrated within the scapulohumeral joint under conditions of complete asepsis.

SUMMARY:
Rotator Cuff Syndrome is a commonly encountered musculoskeletal disorder in clinical practice, with an incidence ranging from 0.3% to 5.5%, and an annual prevalence of 0.5% to 7.4%. In addition, over time, with a monthly rate of 0.26%, this condition can progress to complete rotator cuff tendon injury resulting in worsening pain and shoulder function. The etiology of Rotator Cuff Syndrome is still controversial. What the investigators know is that in tendinopathies there are histological changes in the structure of the tendons, resulting in a change in the mechanical properties of the tendons and leading to a chronic often disabling pain condition. Although conservative therapy should still be considered the first choice in cuff tendinopathies, The clinical results of the various types of nonsurgical treatments are still mixed and often show poor efficacy. This explains the growing interest of the scientific community in developing new biological therapies that can both improve shoulder function and promote tendon healing. The aim of the study is to evaluate, through the Constant Murley Score (CMS), the performance of intra-articular treatment with a collagen-based medical device (MD-Shoulder Collagen Medical Device) in recovering joint function and reducing pain in Rotator Cuff Syndrome.

DETAILED DESCRIPTION:
This is a pilot monocentric Clinical Investigation based on a one sample design. The purpose of this research is to evaluate, through the CMS functional scale, the performance of intra-articular treatment with a collagen-based medical device in recovering joint function and reducing associated pain. The safety of the treatment will also be assessed. Variables will be assessed at 6 different times points: at baseline (day0), after weeks 2, weeks 4, months 3, months 6, and after months 12.

The total duration of the study will be 16 months. There will be a 4-month subject selection and recruitment period and a 12-month treatment and observation period.

A total of 24 subjects with painful shoulder in Rotator Cuff Syndrome will be enrolled. The recruitment phase will be closed no sooner than the number of subjects planned in the study has been reached. Enrollment will involve subjects with rotator cuff syndrome who are eligible according to the selection criteria. Diagnosis will be performed by the Principal Investigator through clinical examination and instrumental investigation with shoulder MRI. The investigators will explain the rationale for the investigation plan and the procedures involved to the eligible subjects. Consent to participate in the study will then be sought. Prior or ongoing the treatments of any kind will be documented.

In order to monitor analgesic consumption (Celecoxib 200mg / Paracetamol 1000 mg) used during the study in case of pain onset, a clinical diary will be given to the subject in which to indicate the day and dose of medication used.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with age > 18 years.
* Subjects with shoulder pain for at least 3 month.
* Subjects with a diagnosis of rotator cuff tendinopathy, subacromial conflict syndrome, partial rotator cuff tendon injuries (injuries A and B according to Snyder's Classification).
* Subjects with a CMS score between 40 and 75.
* Subjects who understood and signed the Informed Consent to Active Participation in the study.
* Subjects able to understand the conditions of the study and participate throughout the duration.

Exclusion Criteria:

* Subjects with complete rotator cuff lesions (C lesions according to Snyder's classification).
* Subjects with shoulder instability.
* Subjects with adhesive retractile capsulitis.
* Subjects undergoing Hyaluronic Acid and/or cortisone infiltration in a period < 3 months.
* Subjects with diabetes mellitus.
* Subjects with uncontrolled thyroid disease.
* Subjects with coagulopathies.
* Subjects on chronic treatment with immunosuppressants.
* Subjects with an allergy to porcine collagen.
* Subjects in pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randelli RP Pietro Simone, Prof, Principal Investigator — Gaetano Pini CTO
Locations (1):
- Gaetano Pini CTO, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- MD-Shoulder Medical Device: MD-Shoulder Medical Device type I collagen based
  MD-Shoulder Collagen Medical Device: Only one experimental group is scheduled by the Investigation Plan to be treated with 2-mL volume ultrasound-guided infiltrations of MD-Shoulder Collagen Medical Device (GUNA, Milan-Italy).
  Subjects will be treated with number one ultrasound-guided infiltration at the time of enrollment, 2 weeks after enrollment, and 4 weeks after enrollment.
  Intra-articular infiltrations will be performed with 5cc syringes and 22-gauge needles.
  MD-Shoulder Collagen Medical Device will be infiltrated within the scapulohumeral joint under conditions of complete asepsis.
Period: Overall Study
Arm/Group | MD-Shoulder Medical Device
Started | 24
Completed | 23
Not Completed | 1
Not completed — withdrawn | 1

BASELINE CHARACTERISTICS:
Arm/Group | MD-Shoulder Medical Device
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Constant-Murley Score (CMS) at 3 Months
Description: The primary outcome is the change from baseline in the Constant-Murley Score (CMS) at 3 months after the first intra-articular injection. The CMS is a validated clinical scale ranging from 0 to 100 points, where higher scores indicate better shoulder function and less pain. It includes four subdomains: pain (15 points), activities of daily living (20 points), range of motion (40 points), and strength (25 points). An increase of at least 13 points is considered very clinically significant. Results will be analyzed as the mean change in CMS from baseline (Day 0) to Month 3.
  Unit of Measure:
  Points on the Constant-Murley Scale (0-100)
Time Frame: 3 months after baseline (Day 0)
Population: A total of 24 subjects with painful shoulder in rotator cuff tendinopathy have been enrolled.
  Only subjects were be included:
  * belonging to the U.O.C. 1st Orthopedic Clinic (Gaetano Pini Orthopedic Institute, Milan, Italy);
  * who meet the inclusion criteria and have no exclusion criteria.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MD-Shoulder Medical Device
Number analyzed (Participants) | 23
units on a scale | 10.03 [3.63 to 16]
Statistical Analysis 1: Comparison: MD-Shoulder Medical Device; Statistical analysis was performed on 23 participants with valid Constant-Murley Score (CMS) data at both baseline and 3-month follow-up; Test type: Other — Paired-sample t-test was used to assess the change in Constant-Murley Score from baseline to 3 months; p = 0.001, t-test, 2 sided; Mean Difference (Net) = 10.03, 95% CI 2-sided [3.63 to 16.00], Standard Error of Mean 2.124 — Mean change from baseline in CMS at 3 months. Higher scores represent better shoulder function. Positive difference indicates clinical improvement

2. Secondary Outcome: Evaluation of MD-Shoulder Collagen Medical Device Performance Using the Constant-Murley Score
Description: Secondary Endpoints will consist of the evaluation of MD-Shoulder Collagen Medical device through CMS at months 6 and months 12 compared to day 0.
Time Frame: months 6, months12
Reporting Status: Not Posted

3. Secondary Outcome: Evaluation of MD-Shoulder Collagen Medical Device With Numeric Rating Scale
Description: Secondary Endpoints will consist of the evaluation of MD-Shoulder Collagen Medical Device, with NRS (Numeric Rating Scale) at weeks 2, weeks 4, months 3, mouth 6, mouth 12 compared to day 0.
Time Frame: weeks 2, weeks 4, months 3, months 6, months 12
Reporting Status: Not Posted

4. Secondary Outcome: Evaluation of MD-Shoulder Collagen Medical Device With American Shoulder and Elbow Surgeons (ASES)Scores Range From 0 to 100 With a Score of 0 Indicating a Worse Shoulder Condition and 100 Indicating a Better Shoulder Condition
Description: Secondary Endpoints will consist of the evaluation of MD-Shoulder Collagen Medical with American Shoulder and Elbow Surgeons (ASES), Simply Shoulder Test (SST) and Range Of Motion (ROM) at months 3, mouth 6, mouth 12 compared to day 0
Time Frame: months 3 months 6, months 12
Reporting Status: Not Posted

5. Secondary Outcome: Evaluation of MD-Shoulder Collagen Medical Device With Simply Shoulder Test (SST), the Items on the Scale Measure the Ability of the Affected Shoulder to Perform Work Duties, Dressing, Bathing, Lifting, Carrying and Throwing.
Description: Secondary Endpoints will consist of the evaluation of MD-Shoulder Collagen Medical Device with simply shoulder test (SST) at months 3, mouth 6, mouth 12 compared to day 0
  number of "yes"/number of completed items 100 = % of "yes" response. 0 = worst and 100 = best function
Time Frame: months 3, months 6, months12
Reporting Status: Not Posted

6. Secondary Outcome: Evaluation of MD-Shoulder Collagen Medical Device With Range of Motion (ROM).
Description: Secondary Endpoints will consist of the evaluation of MD-Shoulder Collagen Medical with Range Of Motion (ROM) at months 3, mouth 6, mouth 12 compared to day 0
Time Frame: months 3, months 6, months12
Reporting Status: Not Posted

7. Secondary Outcome: Evaluation of MD-Shoulder Collagen Medical With Cuff Integrity at Mouth 12 Compared to Day 0 by Performing With Magnetic Resonance Imaging (MRI) of the Treated Shoulder.
Description: Secondary Endpoints will consist of the evaluation of MD-Shoulder Collagen Medical with cuff integrity at mouth 12 compared to day 0 by performing with Magnetic Resonance Imaging (MRI) of the treated shoulder.
Time Frame: month 12
Reporting Status: Not Posted

8. Secondary Outcome: Evaluation of MD-Shoulder Collagen Medical With Assessment of Analgesic Drug Unit Consumption Based on Clinical Diary at Various Phases of the Study.
Description: Secondary Endpoints will consist of the evaluation of MD-Shoulder Collagen Medical with Analgesic consumption at various phases of the study with use of clinical diary
Time Frame: months 3, months 6, months 12
Reporting Status: Not Posted

9. Secondary Outcome: Safety Evaluation
Description: Evaluation of Adverse Events.
Time Frame: weeks 2, weeks 4, months 3, months 6, months 12
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: They were followed for 12 months, constantly monitoring any adverse events During the entire investigation period, the Investigators team reported n°1 Adverse Event (AE) at time T0 after the first infiltration. No serious adverse events (SAEs) occurred in the 24 patients in the 12-month study period.
Description: Adverse events were assessed through non-systematic observation over 12 months. All-cause mortality, serious adverse events, and other adverse events were not systematically assessed, as they were not among the pre-specified study endpoints.
Arm/Group | MD-Shoulder Medical Device
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 1/24
OTHER ADVERSE EVENTS (reported when occurring in more than 4.2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MD-Shoulder Medical Device (N=24)
Local redness following infiltration (General disorders) | 1 (1) — Observed after first injection at time T0.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-15): https://cdn.clinicaltrials.gov/large-docs/84/NCT05489484/Prot_SAP_002.pdf